CLINICAL TRIAL: NCT00651352
Title: A Single Dose Bioequivalence Study of 2mg and 4mg Nicotine Lozenges
Brief Title: A Single Dose Bioequivalence Study OfTwo Formulations Of Nicotine Lozenges
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S3010567
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Volunteer Smokers
Keywords: NRT; Bioequivalence; Nicotine
MeSH Terms: interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 mg nicotine prototype (Experimental): 2 mg nicotine prototype
  Interventions: Drug: 2 mg nicotine prototype
- 2 mg nicotine lozenge (Active Comparator): marketed formulation
  Interventions: Drug: 2 mg nicotine lozenge
- 4 mg nicotine prototype (Experimental): 4 mg
  Interventions: Drug: 4 mg nicotine prototype
- 4 mg nicotine lozenge (Active Comparator): 4 mg
  Interventions: Drug: 4 mg nicotine lozenge

INTERVENTIONS:
Drug: 4 mg nicotine lozenge — marketed formulation
  Other Names: Nicotine
  Arms: 4 mg nicotine lozenge
Drug: 2 mg nicotine lozenge — marketed formulation
  Arms: 2 mg nicotine lozenge
Drug: 2 mg nicotine prototype — 2 mg
  Arms: 2 mg nicotine prototype
Drug: 4 mg nicotine prototype — 4 mg
  Arms: 4 mg nicotine prototype

SUMMARY:
Open label, single dose, four-way crossover in healthy smokers. Each subject will be treated with a single dose or four study treatments in a randomized sequence.

ELIGIBILITY:
Inclusion Criteria:

* Subject is either male or female between 18 - 55 years of age inclusive.
* Subject has a BMI within the range 19-27 kg/m². [BMI = Weight (kg) ÷ Height (m)²].
* Subject admits to having smoked commercially-available cigarettes daily for the preceding 12 months and to routinely smoking his or her first cigarette within 30 minutes upon awakening.
* Subject is in good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities as assessed by medical history, physical examination, electrocardiogram (ECG) and clinical laboratory test results (hematology, biochemistry and urinalysis) are within normal limits.
* If female, subject of childbearing potential is practicing a reliable method of contraception in the opinion of the investigator.
* Subject understands and is willing, able, and likely to comply with all study procedures and restrictions.
* Subject demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent.

Exclusion Criteria:

* If female, subject is pregnant, has a positive serum pregnancy test during screening, or is breast-feeding.
* Subject has a disease or condition that may interfere with the oral absorption of the study drugs.

  1. A medical history that, in the opinion of the investigator, might jeopardize the safety of the subject (e.g. rheumatoid arthritis, circulatory problems, recent myocardial infarction, cerebrovascular accident within 12 weeks prior to first study session, unstable or worsening angina pectoris, Prinzmetal's angina or severe cardiac arrhythmia).
  2. A medical history which, in the opinion of the investigator, might impact the validity of the study results and may require pharmacotherapy or prevent the subject from finishing the study.
  3. Oral surgery within 4 weeks of dosing, dental work or extractions within 2 weeks of dosing, or presence of any clinically significant (as determined by the principal investigator) oral pathology including lesions, sores or inflammation.
* Subject has used chewing tobacco or tobacco products other than cigarettes within 21 days of Visit 1.
* Subject has abused alcohol or other substances within two years of screening. For the purposes of this study, alcohol abuse is defined as daily use of greater than two drinks per day.
* Subject has a positive urine drug screen for cannabinoids, amphetamine, cocaine, ecstasy, methamphetamine, or opiates.
* Subject has a positive serum hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV) test result.
* Subject has known or suspected intolerance or hypersensitivity to any of the study materials or closely related compounds or any of their stated ingredients.
* Subject has a genetic deficiency with an inability to metabolize aspartame or phenylalanine, or has been diagnosed with phenylketonuria.
* Subject has participated in another clinical study or received an investigational drug within 30 days of the first study session or previously participated in this study.
* Subject has donated or experienced significant blood loss within 56 days of Visit 2, donated plasma within 7 days of Visit 2, or has a hemoglobin value of <12.0g/dL.
* Subject has been treated with any known enzyme-altering agents (e.g., barbiturates, phenothiazines, cimetidine, theophyllines) within 30 days prior to the first study session.
* Subject has used any nicotine replacement therapy within 21 days prior to the first study session.
* Subject has used any over-the-counter (OTC) medication or herbal supplements within 48 hours prior to administration of study treatment.
* Subject has used any prescription medication within 14 days prior to each study session, excluding hormonal contraceptive or hormone replacement therapy.
* Subject is a member of the study site staff or an employee of the sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To compare the 2mg prototype lozenge to the 2mg standard lozenge in terms of AUC0-infinity, tmax, t½, and Kel, and likewise 4mg prototype lozenge to 4mg standard lozenge. | 12 hours

SECONDARY OUTCOMES:
• To compare the 2mg prototype lozenge to the 2mg standard lozenge in terms of AUC0-infinity, tmax, t½, and Kel, and likewise with the 4mg prototype lozenge to 4mg standard lozenge; | 12 hours
• To evaluate the safety of the 2mg and 4mg prototype lozenges. | Study period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline